CLINICAL TRIAL: NCT01205074
Title: ¹³C-Methacetin Breath Test (MBT) Methodology Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Meridian Bioscience, Inc. (Industry)
Other Study IDs: METH-EX-610- HMO - CTIL
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Subjects; Chronic Liver Disease; Cirrhosis
Keywords: Patients with chronic liver disease and cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Ethanol

ARMS (6):
- Repeatability (Experimental)
  Interventions: Device: 13C Methacetin Breath Test
- COPD (Experimental)
  Interventions: Device: 13C Methacetin Breath Test
- Smokers (Experimental)
  Interventions: Device: 13C Methacetin Breath Test
- CYP450 1A2 Inhibitors (Experimental)
  Interventions: Device: 13C Methacetin Breath Test; Dietary Supplement: Grape fruit juice
- Cirrhosis Beta Blockers (Experimental)
  Interventions: Device: 13C Methacetin Breath Test; Drug: Non selective beta blocker - Propranolol
- Alcohol (Experimental)
  Interventions: Device: 13C Methacetin Breath Test; Dietary Supplement: Ethanol

INTERVENTIONS:
Device: 13C Methacetin Breath Test
Dietary Supplement: Grape fruit juice
  Arms: CYP450 1A2 Inhibitors
Drug: Non selective beta blocker - Propranolol
  Arms: Cirrhosis Beta Blockers
Dietary Supplement: Ethanol
  Arms: Alcohol

SUMMARY:
Several factors will be tested to see if they have an influence on the methacetin breath test results. Each one of the factors has been raised as a possible source of distortion of the MBT result.

I. Variability between same tests on same subject MBT. Repeatability will be tested in both healthy individuals and patients with chronic liver disease.

II. COPD - Chronic obstructive pulmonary disease is a leading cause of death worldwide, and can potentially have an effect on the MBT since the breath test is based on CO2 production and these subjects may have abnormal CO2 production.

III. Smoking- 13C Methacetin is metabolized by healthy hepatocytes reflecting hepatic microsomal function of CYP1A2, and smoking may cause induction of CYP1A2. Furthermore, internal preliminary data has shown signs that there is an influence of smoking on the MBT ranges.

IV. Age- Empirical data on several hundred subjects with chronic liver disease has shown that age is a significant factor in determining the probability of disease severity and preliminary data in normal subjects have shown changes in MBT with age.. Therefore, the effect of age has to be elucidated in an orderly fashion.

V. CYP450 1A2 Inhibitors- Several drugs and food items inhibit CYP450 1A2 and may affect the MBT.

VI. Alcohol - Alcohol ingestion leads to induction of hepatic CYP and at a later stage to inhibition due to liver damage. Acute alcohol ingestion may therefore effect MBT results.

VII. Beta-blockers - beta blocker are affecting portal hypertension and may affect hepatic blood flow and thereby the outcome of the methacetin breath test.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - General

* Adult subjects with 18 years of age or older
* Women of childbearing potential must have a negative serum or urinary hCG pregnancy test within 7 days prior to enrollment. During the study these women must use 2 methods of contraception.
* Subject has given written informed consent, prior to any study related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn at any time without prejudice to future medical care.

Exclusion Criteria - General

* Severe heart, pulmonary or renal disease.
* Patient has previous surgical bypass surgery for morbid obesity
* Patient has extensive small bowel resection
* Any major surgery in the past 3 months.
* Patient is a recipient of any organ transplant
* Pregnant or breastfeeding women.
* Patient allergic to acetaminophen
* Patients who are taking hepatotoxic drugs
* Patient, based on the opinion of the investigator, should not be enrolled into this study.
* Patients unable or unwilling to sign informed consent
* Patients that are participating in other clinical trials evaluating experimental treatments or procedures or have participated in a clinical trial in the past 3 months.

Exclusion Criteria (Day of MBT-general)

* Patient has not fasted for 8 hours.
* Patient has smoked on the day of the test.
* Patient that has taken drugs that can interfere with methacetin metabolism: fluvoxamine, amiodarone, ciprofloxacin, cimetidine, rifampin, carbamazepine within the last 24 hours.
* Patient has taken Tylenol or any other acetaminophen related medications within the past 24 hours.
* Patients that received any new medication in the last 48 hours.
* Patients that still suffer from any previous clinical intervention (e.g. biopsy)
* Have not consumed alcohol 24 hours prior the MBT and not consume on a regular basis more than 40gr for male and 20gr for female per day.

Inclusion Criteria (Repeatability):

Healthy Subjects:

* No known liver disease
* Non smokers
* BMI =20-25 kg/m2
* Normal liver enzymes (ALT < 40 U/L for men, < 30 U/L for women)
* Not taking any medications
* No known on-going chronic medical conditions (apart from allergy or orthopaedic conditions not requiring chronic therapy).
* Normal abdominal ultrasound (US)

Cirrhotics:

* Diagnosis of cirrhosis by liver biopsy
* Or strong suspicion of cirrhosis by accepted criteria for the clinical diagnosis of cirrhosis (e.g. peripheral edema or varices, palpable hard left lobe of the liver, small right lobe span or palpable splenomegaly), and/or radiological evidence of cirrhosis (by abdominal sonography, computer assisted axial tomography, or magnetic resonance imaging, showing a nodular liver and/or portosystemic collaterals with portal vein patency and/or ascites and/or splenomegaly, and/or colloid shift on a colloid-isotope liver-spleen scan), and/or laboratory variables (platelets <100,000/mm3, albumin< 3.5g/dL, or INR >1.3)

Chronic Liver Patient (non cirrhotic):

Patient who has been diagnosed with chronic liver disease for more than 6 months.

Inclusion Criteria (COPD):

* No known liver disease
* BMI 20- 25 kg/m2
* Normal liver enzymes (ALT < 40 U/L for men, < 30 U/L for women)
* Patients with a COPD exacerbation with elevated PCO2 levels (> 50 mmHg)
* Without clinically overt right heart failure
* Ceased smoking for at least one month
* No other overt clinical dysfunction of major organ system

Inclusion criteria (Smoker):

Smokers:

* No known liver disease
* Active smoker of at least 10 cigarettes/day (stable number of cigarettes during past month - not currently trying to quit).
* BMI 20- 25 kg/m2
* Normal liver enzymes (ALT < 40 U/L for men, < 30 U/L for women)
* Not taking any medications
* No known chronic medical conditions

Inclusion criteria (CYP450 1A2 inhibitors):

Healthy Subjects:

* No known liver disease
* Non smokers
* BMI 20- 25 kg/m2
* Normal liver enzymes (ALT < 40 U/L for men, < 30 U/L for women)
* Not taking any medications
* No known chronic medical conditions (allergy or orthopaedic condition not requiring chronic therapy allowed).
* Normal abdominal US

Cirrhotic subjects:

* Diagnosis of cirrhosis by liver biopsy
* Or strong suspicion of cirrhosis by accepted criteria for the clinical diagnosis of cirrhosis (e.g. peripheral edema or varices, palpable hard left lobe of the liver, small right lobe span or palpable splenomegaly), and/or radiological evidence of cirrhosis (by abdominal sonography, computer assisted axial tomography, or magnetic resonance imaging, showing a nodular liver and/or portosystemic collaterals with portal vein patency and/or ascites and/or splenomegaly, and/or colloid shift on a colloid-isotope liver-spleen scan), and/or laboratory variables (platelets <100,000/mm3, albumin< 3.5g/dL, or INR >1.3)
* Not receiving medication which is metabolized by CYP450 1A2

Inclusion criteria (Beta Blockers):

* Diagnosis of cirrhosis (by liver biopsy or clinical diagnosis):

Strong suspicion of cirrhosis by accepted criteria for the clinical diagnosis of cirrhosis (e.g. peripheral edema or varices, palpable hard left lobe of the liver, small right lobe span or palpable splenomegaly), and/or radiological evidence of cirrhosis (by abdominal sonography, computer assisted axial tomography, or magnetic resonance imaging, showing a nodular liver and/or portosystemic collaterals with portal vein patency and/or ascites and/or splenomegaly, and/or colloid shift on a colloid-isotope liver-spleen scan), and/or laboratory variables (platelets <100,000/mm3, albumin< 3.5g/dL, or INR >1.3)

* Naive to Beta Blockers - with a clinical indication for initiating therapy (eg. esophageal varices, portal hypertensive gastropathy)
* Resting pulse > 60 beats per minute
* Non smoker

Inclusion criteria (Alcohol):

* No known liver disease
* Non smokers
* BMI 20- 25 kg/m2
* Normal liver enzymes (ALT < 40 U/L for men, < 30 U/L for women)
* Not taking any medications
* No known chronic medical conditions. (Allergy or orthopaedic condition not requiring chronic therapy allowed).
* Normal abdominal US

Exclusion Criteria:

General

* Severe heart, pulmonary or renal disease.
* Patient has previous surgical bypass surgery for morbid obesity
* Patient has extensive small bowel resection
* Any major surgery in the past 3 months.
* Patient is a recipient of any organ transplant
* Pregnant or breastfeeding women.
* Patient allergic to acetaminophen
* Patients who are taking hepatotoxic drugs
* Patient, based on the opinion of the investigator, should not be enrolled into this study.
* Patients unable or unwilling to sign informed consent
* Patients that are participating in other clinical trials evaluating experimental treatments or procedures or have participated in a clinical trial in the past 3 months.

Exclusion Criteria (Day of MBT-general)

* Patient has not fasted for 8 hours.
* Patient has smoked on the day of the test.
* Patient that has taken drugs that can interfere with methacetin metabolism: fluvoxamine, amiodarone, ciprofloxacin, cimetidine, rifampin, carbamazepine within the last 24 hours.
* Patient has taken Tylenol or any other acetaminophen related medications within the past 24 hours.
* Patients that received any new medication in the last 48 hours.
* Patients that still suffer from any previous clinical intervention (e.g. -
* Have not consumed alcohol 24 hours prior the MBT and not consume on a regular basis more than 40gr for male and 20gr for female per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit Hadassah Medical Center, Jerusalem, Israel